CLINICAL TRIAL: NCT04184063
Title: A Pilot Exploratory, Randomised, Placebo-controlled, Double Blinded, Cross-over , Phase 2a Study to Explore Efficacy and Safety of NBMI Treatment in Patients With Progressive Supranuclear Palsy (PSP) or Multiple System Atrophy (MSA)
Brief Title: Study of NBMI Treatment in Patients With Atypical Parkinsons (PSP or MSA)
Acronym: EMERA006
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EmeraMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: EMERA006
Record Dates: First submitted 2019-07-29; First posted 2019-12-03 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Progressive Supranuclear Palsy; Multiple System Atrophy
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Multiple System Atrophy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active treatment with NBMI (Experimental)
  Interventions: Drug: NBMI
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: NBMI — NBMI active treatment
  Arms: active treatment with NBMI
Other: Placebo — Placebo for comparison
  Arms: Placebo

SUMMARY:
In total 20 subjects will be enrolled at one participating site -UMC Ljubljana. The 20 subjects will be treated with placebo and NBMI 300 mg in a cross-over design. In case of subject drop-outs, additional subjects may be enrolled as decided by the Sponsor, to allow for expected number of evaluable subjects in each group.

DETAILED DESCRIPTION:
· The study's primary objective is: To explore the efficacy of 28 days NBMI treatment on motor and non-motor symptoms and heath related quality of life in patients with Progressive Supranuclear Palsy or Multiple Systems Atrophy disease.

The study's secondary objectives are:

* to explore safety and tolerability of 28 day NBMI treatment in patients with Progressive Supranuclear Palsy or Multiple Systems Atrophy.
* to investigate the efficacy of NBMI daily oral administration for 28 days on fatigue in MSA and PSP patients,
* to investigate the efficacy of NBMI daily oral administration for 28 days on depression in MSA and PSP patients.

The study's exploratory aims are:

* to explore the effect of NBMI treatment on patient's brain iron levels as evaluated by MRI imaging,
* to explore the effect of NBMI on brain metabolism with FDG- PET- CT brain imaging,
* to explore the pharmacokinetics of NBMI in patients with PSP or MSA.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has clinically confirmed documented diagnosis of PSP or MSA, according to the current clinical criteria.
2. Patient has a brain MRI finding consistent with the diagnosis of PSP or MSA at Screening.
3. Patient is aged 40 years to 85 years inclusive at screening age.
4. Patient is fluent in the local language and possesses sufficient auditory and visual capacities to allow neuropsychological testing.
5. Patient and caregiver are able to read and understand informed consent.
6. Patient is on a stable therapy for PSP, MSA for at least 1 month prior to screening visit.
7. If the patient received i.v. amantadine treatment, the last infusion must have been administered at least 6 months prior to the screening (V01).
8. Availability of a caregiver who sufficiently knows the patient and will be able to accompany the patient on the study visits and to participate in study assessments of the patient where required.
9. Female patients are only eligible for the study if they are either surgically sterile or at least 2 years postmenopausal or have a negative result of serum hCG test at screening and apply to criteria no. 10.
10. Female of childbearing potential can only participate in the study if willing to use acceptable, effective methods of contraception during the trial and for three month after the end of trial participation as defined in point 6.7. of this protocol.
11. Male patients must either be surgically sterile or he and his female spouse/partner who is of childbearing potential must be willing to use highly effective methods of contraception consisting of 2 forms of birth control (1 of which must be a barrier method) starting at screening and continuing throughout the study.
12. Patient provides written informed consent.

Exclusion Criteria:

1. Known history or presence of clinically significant other neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, genitourinary, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results.
2. Known or suspected allergy hypersensitivity or idiosyncratic reaction to NBMI or any other drug substances with similar activity.
3. Patient has known contraindication for MRI imaging such as MRI-incompatible metallic endoprosthesis or MRI-incompatible stent implantation or other as judged by the Investigator.
4. Patient has claustrophobia that could prevent MRI imaging
5. History of drug or alcohol addiction requiring treatment.
6. Patient who had previous chronic exposure (within one year before recruitment) to iron from taking preparations/medications for rising iron
7. History of malabsorption within the last year or presence of clinically significant gastrointestinal disease or surgery that may affect drug bioavailability, including but not limited to cholecystectomy.
8. Patient is ridden to bed.
9. Presence of hepatic or renal dysfunction. (SGOT and SGPT and bilirubin > X2 UNL. creatinine > 1.5mg/dl)
10. Female patient who is pregnant (serum hCG level consistent with pregnancy diagnosis); or breastfeeding.
11. Participation in a clinical trial that involved administration of an investigational medicinal product within 90 days prior to drug administration, or recent participation in a clinical investigation that, in the opinion of the Investigator, would jeopardize subject safety or the integrity of the study results.
12. Patient has a history with evidence of cerebrovascular disease (ischemic or haemorrhagic), or diagnosis of possible, probable or definite vascular Parkinsonism or dementia.
13. Have clinically significant abnormal laboratory values (e.g. liver enzymes)
14. Have clinically significant findings from a physical examination (e.g. fever)
15. Patient has claustrophobia that could prevent him from attending MRI imaging

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Changes in Progressive Supranuclear Palsy rating Scale (PSPRS) individual scales scores from baseline in PSP patients compared to placebo treatment | through study completion, an average of 85 days
  For PSP specific scales (to study on PSP patients):- Progressive Supranuclear Palsy rating Scale is used as a quantitative measurement of disability in PSP patients. The available total score ranges from 0 (normal) to 100. Six items are rated on a 3-point scale (0-2) and 22 are rated on a 5-point scale (0-4). The History/Daily Activities area includes seven items with a total maximum of 24 points, the mentation area four items with 16 points, the bulbar area two items with 8 points, the ocular motor area four items with 16 points, the limb motor area six items with 16 points and the gait area five items with 20 points. Scores from each subscale is summed and combined to compute a total score. Higher values for each scale range provided represent worse outcome.
Changes in FAB individual scales scores from baseline in PSP patients compared to placebo treatment | through study completion, an average of 85 days
  For PSP specific scales (to study on PSP patients):- Frontal Assessment Battery (FAB) is a brief tool that can be used at the bedside or in a clinic setting to assist in discriminating between dementias with a frontal dysexecutive phenotype and Dementia of Alzheimer's Type (DAT). The FAB has validity in distinguishing Fronto-temporal type dementia from DAT in mildly demented patients (MMSE > 24). The 6 subtests of the FAB explore the following: conceptualization and abstract reasoning; mental flexibility; motor programming and executive control of action; resistance to interference; inhibitory control; and environmental autonomy. Each subtest is scored from 3 (better score) to 0, for a maximum score of 18. Scores from each subscale is summed and combined to compute a total score. Higher scores indicate better performance.
Changes in Unified Multiple System Atrophy Rating Scale (UMSARS) individual scale from baseline in MSA patients compared to placebo treatment | through study completion, an average of 85 days
  Unified Multiple System Atrophy Rating Scale (UMSARS) is a multimodal scale used to provide a surrogate measure of disease progression in multiple system atrophy. Components: Part I, historical, 12 items; Part II, motor examination, 14 items; Part III, autonomic examination (descriptive); and Part IV, global disability scale. Scale is used by physician who rates the average functional situation for the past 2 weeks (unless specified) according to the patient and caregiver interview. Scores are ranging from 0 to 104; higher scores indicate greater impairment. Rating scale includes autonomic symptoms (questions 9-12 - activities of daily living subscale [range 0-16]) and motor symptoms (questions 1-8 - activities of daily living subscale [range 0-32] and the UMSARS motor examination subscale, range 0-56), as well as their effect on activities of daily life (activities of daily living subscale, range 0-48). Scores from each subscale is summed and combined to compute a total score.
Changes in Non-Motor Symptoms assessment scale (NMSS) individual scale from baseline in MSA patients compared to placebo treatment | through study completion, an average of 85 days
  Non-Motor Symptoms assessment scale for Parkinson s disease assesses 9 domains: Cardiovascular (2 items); Sleep/fatigue (4 items); Mood/cognition (6 items); Perceptual problems/hallucinations (3 items); Attention/memory (3 items); Gastrointestinal tract (3 items); Urinary function (3 items); Sexual function (2 items); and Miscellaneous (4 items). Score for each item is based on a multiple of severity (from 0 to 3) and frequency scores (from 1 to 4). The scale can therefore capture symptoms that are severe but relatively infrequent and those that may be less severe but persistent. Scores from each subscale is summed and combined to compute a total score. Lower result indicates better health results.
Changes in QOL individual scores from baseline by MSA questionnaire in MSA patients | through study completion, an average of 85 days
  MSA-QoL is a patient-rated health-related Quality of life scale for patients with multiple system atrophy (MSA). It is designed to test its psychometric properties. Items are given a standard five response option format (0 - no problem to 4 - extreme problem), where higher scores indicate worse health results. The available total score ranges from 0 to 160 (there are 40 questions altogether).
Changes in QOL individual scores from baseline by MSA questionnaire in MSA patients using Visual Analog score | through study completion, an average of 85 days
  MSA-QoL is a patient-rated health-related Quality of life scale for patients with multiple system atrophy (MSA). Visual Analog score is designed to determine overall life satisfaction in patient with MSA. Scale is given response option format (0 - extremely unsatisfied with life 100 - extremely satisfied with life), where higher scores indicate better satisfaction/quality of life.
Changes in QOL individual scores from baseline by EQ-5D score in PSP patients compared to placebo treatment | through study completion, an average of 85 days
  EuroQol (EQ-5D) is a standard Health related Quality of questionnaire scale that is completed by patient. It comprises from questions related to 5 different aspects of health such as mobility, self- care, usual activities, pain/ discomfort, anxiety/depression) and a visual health assessment scale completed by patient graphically. Visual scale has following range: 0 (worst possible state) - 100 (best possible state). A scale is completed by patients.

SECONDARY OUTCOMES:
Changes in Parkinson's Disease Fatigue Score (PFS) score from Baseline - V1 to V2 (D29) and V1 to V5 (D57) in PSP and MSA patients compared to placebo treatment | through study completion, an average of 85 days
  Parkinson's Disease Fatigue Score (PFS) is a fatigue rating scale that comprises from series of statements (16) about fatigue and the impact that it can have. Patients are asked to indicate how well the statements describe their feelings and experiences over the past two weeks. Maximal number of points is 80, lower results are indicating better health.
Changes in Beck's Depression Inventory (BDI) scale (MSA patients) score from Baseline V1 to V2 (D29) and to V4 (D57) compared to placebo treatment | through study completion, an average of 85 days
  In MSA patients Beck's Depression Inventory will be used as a measure of depression in MSA patients. It is a patient reported scale.
  Confidential: The information in this study protocol is legally privileged and confidential. Any disclosure, copying or distribution of the information contained within is strictly prohibited without written authorization from EmeraMed Ltd.
  lower end indicate normal status. A maximum achievable score is 15, the cut off between depressed and not depressed subjects is around the score 5.
Changes in Geriatric depression scale (GDS) (PSP patients) score from Baseline - V1 to V2 (D29) and to V4 (D57) compared to placebo treatment | through study completion, an average of 85 days
  GDS is a 15-item self reported assessment tool designated to identify depression in the elderly, frequently used in clinical practise and research. Scale is completed by patients. The subjects answers questions with Yes or No, and the answers are scored by 0 and 1, respectively.
  Confidential: The information in this study protocol is legally privileged and confidential. Any disclosure, copying or distribution of the information contained within is strictly prohibited without written authorization from EmeraMed Ltd.
  lower end indicate normal status. A maximum achievable score is 15, the cut off between depressed and not depressed subjects is around the score 5.
Frequency, type and severity of adverse events compared to placebo treatment . | through study completion, an average of 85 days
  Adverse Events (AEs) will be reported throughout the study. AEs will be classified as treatment - emergent adverse events if their start lies after the first dose of IMP and before End of the study or Early Discontinuation visit. AEs will be coded according to MeDRA (Medical Dictionary for Regulatory Activities), latest version. They will be tabulated, summarised and divided by treatment group. AEs tabulation will be done in descending order by event frequency per system organ class. Change from baseline will be calculated for laboratory values and vital signs. Safety clinical chemistry and haematology data that are below lower limit of quantification (LLOQ) will be treated as 50 % of the lower limit value.
Percentage of NBMI-treated patients who develop a response to NBMI. | through study completion, an average of 85 days
  Response will be defined as a change from baseline in any scale for more than 20 % or change for at least one category unit.

OTHER OUTCOMES:
Changes from baseline in brain metabolism as evaluated with Fluorodeoxyglucose Positron Emission Tomography (FDG PET) CT brain imaging compared to placebo treatment | through study completion, an average of 85 days
  Changes from baseline in brain metabolism as evaluated with FDG PET CT brain imaging compared to placebo treatment
Changes from baseline in brain iron levels as detected with Magnetic Resonance Imaging (MRI) imaging methods compared to placebo treatment | through study completion, an average of 85 days
  Changes from baseline in brain iron levels as detected with MRI imaging methods
Pharmacokinetic parameters derived from plasma concentrations of NBMI: Maximum Plasma Concentration [Cmax] | Day 56, 57
  Maximum Plasma Concentration [Cmax]Maximum drug concentration in the samples matrix obtained directly from the observed concentration versus time data.
Pharmacokinetic parameters derived from plasma concentrations of NBMI: AUC0-t | Day 56, 57
  Area Under the Curve [AUC) The area under the plasma concentration-time curve from time-zero to the time of the last quantifiable concentration; calculated using the linear trapezoidal rule.
Pharmacokinetic parameters derived from plasma concentrations of NBMI: AUC0-∞ | Day 56, 57
  Area Under the Curve [AUC)Area under the concentration-time curve from time-zero extrapolated to infinity calculated as AUC0-t + Clast/ λz.
Pharmacokinetic parameters derived from plasma concentrations of NBMI: AUC%Extrap,obs | Day 56, 57
  Area Under the Curve [AUC)The residual area in percentage will be determined by the formula, [(AUC0-∞ - AUC0-t) / AUC0-∞] x 100.
Pharmacokinetic parameters derived from plasma concentrations of NBMI: t1/2 | Day 56, 57
  Apparent terminal elimination half-life (h) determined as: ln2/ λz.
Pharmacokinetic parameters derived from plasma concentrations of NBMI: λz | Day 56, 57
  The terminal elimination rate constant; calculated using linear regression on the terminal portion of the plasma concentration versus time curve.
Pharmacokinetic parameters derived from plasma concentrations of NBMI: T max | Day 56, 57
  Time of maximum analyte concentration (h), obtained directly.

CONTACTS AND LOCATIONS:
Overall Officials: Tanja Turk, M. Pharm, Study Director — CRS d.o.o.
Locations (1):
- Ukc Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No